CLINICAL TRIAL: NCT06543251
Title: The Effects of Training Between High-Intensity Interval and Moderate Continuous Exercise on Respiratory Function and Rhinitis Symptoms in Patients With Allergic Rhinitis.
Brief Title: Effect of High Intensity Interval Exercise Training in Patients With Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wannaporn Tongtako, Ph.D., Principal investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EX PHYSIO SPSC 11
Record Dates: First submitted 2024-08-04; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis; Aerobic exercise; High intensity interval training; pulmonary function; cytokines
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity interval training group (HIIT) (Experimental): the group with high-intensity interval training at a ratio of 1:2 (HIIT) 3 days per week, over a total period of 12 weeks.
  Interventions: Other: High-intensity interval training group (HIIT)
- Moderate continuous training group (MCT) (Experimental): the group with moderate continuous training, 3 days per week, over a total period of 12 weeks.
  Interventions: Other: Moderate continuous training group (MCT)
- Sedentary control group (CON) (Other)
  Interventions: Other: Sedentary control group (CON)

INTERVENTIONS:
Other: High-intensity interval training group (HIIT) — The participants performed HIIT programs for 12 weeks involving walking/running on a treadmill preceded by a 10-min warm-up at low intensity and exercise with high intensity for 1 min at 85%-90% of the maximum heart rate alternating with low intensity at 50%-55% of the maximum heart rate for 2 min, for 24 minutes, and 10-min cool down.
  Arms: High-intensity interval training group (HIIT)
Other: Moderate continuous training group (MCT) — Subject participating in 30-min sessions for 12 weeks and Each session consisted of a 10-min warm up, walking/running on a treadmill 30 minutes at 65-70% Maximum Heart rate and 10-min cool down.
  Arms: Moderate continuous training group (MCT)
Other: Sedentary control group (CON) — The control group had normal daily life.
  Arms: Sedentary control group (CON)

SUMMARY:
The objective of this study was to compare the effects of training between high-intensity interval training and moderate continuous exercise training on the pulmonary function, respiratory muscle strength, symptoms of patients with allergic rhinitis, cytokines, and oxidative stress in patients with allergic rhinitis.

DETAILED DESCRIPTION:
36 patients with allergic rhinitis were divided into 3 groups, 12 people per group: the control group (CON), the group with high-intensity interval training at a ratio of 1:2 (HIIT) and the group with moderate continuous training (MCT), 3 days per week, over a total period of 12 weeks. Before and after the experiment, lung function, respiratory muscle strength, allergic rhinitis symptoms, nasal blood flow rate, peak nasal inspiratory flow, nitric oxide levels, cytokines and quality of life were measured and used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* A patient with allergic rhinitis who underwent a skin prick test and received a positive result.
* Patients with persistent allergic rhinitis, male and female, with symptoms of nasal congestion, sneezing, nasal itching, and runny nose for more than 4 days per week, and an average score of 7 or more in the past week using the allergic rhinitis symptom assessment questionnaire.
* stopped taking all medicine before the study such as antihistamine for 3 days, oral steroid and nasal steroid for at least 2 weeks and leukotriene receptor antagonist for at least a week prior to the study
* had no exercise program, non-smoking and without any food supplementation for at least 6 months prior to the start of the study
* Must not have other respiratory diseases such as bronchitis, pertussis, pneumonia, pneumonitis, aspergilloma, tuberculosis, asthma, lung cancer, emphysema, etc.
* Have a body mass index (BMI) between 18.5 and 24.9 kg/m².
* Complete the Physical Activity Readiness Questionnaire (PAR-Q+) by answering "no" to all questions.

Exclusion Criteria:

* There is an unforeseen circumstance, such as an illness, that prevents participation in the research.
* Less than 80% of the research was completed.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Rhinitis symptom scores | Change from Baseline Rhinitis symptom scores at 12 weeks.
  Nasal symptoms were assessed using Total Nasal Symptom Score (TNSS) questionnaire. The subjects were asked to score symptoms of persistent allergic rhinitis before and after yoga training protocol. The total nasal symptom scores were computed as the sum of four individual nasal symptom scores; nasal congestion, itching, sneezing, and rhinorrhea. The scores ranged from 0 to 3 scale (0=none, 1=mild, 2=moderate, 3= severe)
Peak nasal inspiratory flow | Change from Baseline Peak nasal inspiratory flow scores at 12 weeks.
  The subjects placed a mask, which is turned onto a plastic cylinder through which the air passes during inspiration, over the nose and mouth and inspired forcefully through the nose, with lips tightly closed. Inside the cylinder, there is a diaphragm that moves to the airflow, and the maximum peak flow is registered in a scale range from 30-370 L/min. During the procedure, the subjects placed a mask over the nose and mouth and inspired forcefully through the nose, with lips tightly closed.
Nasal blood flow | Change from Baseline Nasal blood flow scores at 12 weeks.
  Laser Doppler flowmetry (DRT4 moor instrument, UK.) was used to measure of the nasal blood flow (NBF). Before the test each subject rested for one hour in a separate room. During the test, they were instructed to breathe normally breathe and not to speak, cough, or move. A lateral endoscopic probe with a flexible nylon sheath 1.34-mm-diameter flexible nylon sheath was placed to the front of the nose.
Pulmonary Functions | Change from Baseline Pulmonary Functions at 12 weeks.
  The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration.
Respiratory muscle strength | Change from Baseline Respiratory muscle strength at 12 weeks.
  Respiratory muscle strength was assessed by measuring Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) in cmH2O. The participants were in a sitting position using a portable handheld mouth pressure meter (i.e., MicroRPM) with a nose clip. For the MIP measurement, the participants were asked to exhale until they felt no air remaining in their lungs (starting with the functional residual capacity [FRC] point), then held the device on their mouth and inhaled forcefully for 1-2 seconds. For the MEP measurement, the participants were asked to inhale until their lungs were completely filled with air (starting with the total lung capacity [TLC] point), then they kept the device on their mouth and exhaled forcefully for 1-2 seconds
Fraction exhaled nitric oxide | Change from Baseline Fraction exhaled nitric oxide at 12 weeks.
  Participants inhaled deeply for two to three seconds before exhaling slowly. Normally, it took 10 seconds to exhale.
Aerobic capacity | Change from Baseline Aerobic capacity at 12 weeks.
  Aerobic capacity variables were measured by determining maximum oxygen uptake (VO2max) using the Bruce protocol. The subjects ran on a treadmill. At the beginning of the test, the baseline or resting value was collected for the first 3 minutes. The initial speed was set at step 1 (minutes 0-3) at a speed of 1.7 mph with a 10% incline. The test was incremented every 3 minutes. Step 2 (minutes 4-6) was conducted at a speed of 2.5 mph with a 2% incline. The test continued until the subjects could not run any further. Following this, the subjects were cooled down for 3 minutes. The maximum oxygen uptake was measured in milliliters per kilogram per minute (ml/kg/min).

SECONDARY OUTCOMES:
Cytokine in nasal secretion | Change from Baseline Cytokine in nasal secretion at 12 weeks.
  Nasal secretions collection was performed bilaterally with filter paper strips (7x30 mm Whatman No.42, Whatman, Clifton, NJ). Three filter paper strips were sequentially placed on each anterior portion of the inferior turbinate for 10 min. This filter paper strips were collected into appropriate tubes and centrifuged at 3,000 rpm for 5 min at 4 °C and immediately frozen at -70 °C until later analysis.The levels of cytokines were determined by using Sandwich ELISA technique
Rhinoconjunctivitis quality of life questionnaire - 36; Rcq-36 | Change from Baseline quality of life at 12 weeks.
  The quality of life of individuals with allergic rhinitis was assessed using the Rhinoconjunctivitis Quality of Life Questionnaire (Rcq-36). The researcher distributed the questionnaire and asked the participants to fill it out themselves.

CONTACTS AND LOCATIONS:
Overall Officials: Wannaporn Tongtako, Ph.D., Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No